CLINICAL TRIAL: NCT00741624
Title: Mitigating Pain Following Refractive Surgery
Brief Title: Pain Reduce Following Refractive Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FORSIGHT Vision3 (Industry)
Responsible Party: Yair Alster, Forsignt Vision
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0165
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Pain
Keywords: refractive surgery
MeSH Terms: conditions — Pain | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): bilateral post refractive surgery subject
  Interventions: Other: Bandage

INTERVENTIONS:
Other: Bandage — one application for one week

SUMMARY:
applying a material over the exposed stromal bed following refractive surgery to prevent local abrasion and significantly reduce pain

DETAILED DESCRIPTION:
Assessed for pain at 1, 2 and 4 hours and 1, 3 and 5 days. Comparison to non study eye will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent bilateral PRK for myopic correction.
2. Age 18-60.
3. Patient complains of significant pain.
4. Patients able to understand the requirements of the study and willing to follow study instructions, to provide written informed consent to participate, and who agree to comply with all study requirements, including the required study follow-up visits

Exclusion Criteria:

1. Any other anterior segment abnormality other than that associated with PRK.
2. Any abnormalities associated with the eye lids.
3. Prior laser treatment of the retina.
4. Any ophthalmic surgery performed within three (3) months prior to study excluding PRK.
5. Diagnosis of glaucoma.
6. Active diabetic retinopathy.
7. Clinically significant inflammation or infection within six (6) months prior to study.
8. Uncontrolled systemic disease (e.g., diabetes, hypertension, etc.) in the opinion of the Investigator.
9. Participation in any study involving an investigational drug within the past 30 calendar days, or ongoing participation in a study with an investigational device.
10. Specifically known intolerance or hypersensitivity to contact lenses.
11. A medical condition, serious intercurrent illness, or extenuating circumstance that would significantly decrease study compliance, including all prescribed follow-up.
12. Any condition that, in the opinion of the investigator, would jeopardize the safety of the patient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain relief | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: David Verssano, Principal Investigator — Sorasky Medical Center
Locations (1):
- Sorasky Medical Center, Tel Aviv, Israel